CLINICAL TRIAL: NCT02252965
Title: CONSENT - Comparison of metfOrmin XR to IR as moNotherapy in the Newly diagnoSed Type 2 diabEtes Patients for the gastroiNtestinal Tolerability and Efficacy: a Randomized, Parallel Control, Open-label and Multicenter Study
Brief Title: Metformin Extended Release Versus Metformin Immediate Release in Subjects With Type 2 Diabetes
Acronym: CONSENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200084-513
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Results first posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Metformin XR; Metformin IR
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin IR (Active Comparator)
  Interventions: Drug: Metformin IR
- Metformin XR (Experimental)
  Interventions: Drug: Metformin XR

INTERVENTIONS:
Drug: Metformin IR — Subjects will receive Metformin Immediate Release (IR) tablets, orally once daily at a dose of 500 milligram (mg) for 1 week, and then dose will increase with increments of 500 mg every week in first 2 weeks to 1500 mg. After that dose will increase up to maximum dose of 2000 mg for the next 2 weeks and will be maintained at 2000 mg until Week 16.
  Other Names: Glucophage IR
  Arms: Metformin IR
Drug: Metformin XR — Subjects will receive Metformin Extended Release (XR) tablets, orally once daily at a dose of 500 mg for 1 week, and then dose will increase with increments of 500 mg every week in first 2 weeks to 1500 mg. After that dose will increase up to maximum dose of 2000 mg for the next 2 weeks and will be maintained at 2000 mg until Week 16.
  Other Names: Glucophage XR
  Arms: Metformin XR

SUMMARY:
This is a Phase 4, prospective, open label, randomized, parallel controlled multicenter trial in which metformin extended release (XR) will be compared with metformin immediate release (IR) for the gastrointestinal tolerability and efficacy in the newly diagnosed subjects with Type 2 diabetes who have glycosylated hemoglobin (HbA1c) value between 7.0 to 10.0 percent (%).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of Type 2 diabetes mellitus before the screening visit based on the World Health Organization (WHO) diagnostic and classification criteria
* HbA1c value of 7.0-10.0%, inclusive
* Age ranging from 18 to 79 years, inclusive
* Treatment-naive for oral antidiabetic agents (that is, had not received antidiabetic medication previously, or had received antidiabetic medication for at least 14 days and not within 1 month of enrolment)
* Male, or non-pregnant, non-breastfeeding females
* Body mass index (BMI) greater than or equal to (>=) 18.5 and less than (<) 35 kilogram per square meter (kg/m^2)
* In the opinion of the investigator, subjects are well-motivated, capable and willing to continue the study treatment as required during the whole study period, maintain a study dietary, as required for this protocol, attend scheduled visits and be willing to receive phone calls between visits, avoid pregnancy by using an adequate method of contraception throughout the duration of the study for the female subjects of child bearing potential (and if appropriate male subjects with female partners of childbearing potential)
* Written informed consent given before any trial-related activities are carried out

Exclusion criteria:

* Type 1 diabetes
* Previous treatment with insulin or other antidiabetics (including Chinese traditional medicine) for more than 14 days continuously or within 1 month of enrolment
* Any of the protocol-specified cardiovascular conditions within 3 months prior to the screening visit
* Impaired liver function as defined in the protocol
* Serum creatinine values as specified in the protocol
* Known proliferative retinopathy or maculopathy requiring acute treatment, or recurrent major hypoglycemia or hypoglycemic unawareness as judged by the investigator
* Persistent uncontrolled hypertension
* Severe chronic gastrointestinal disease
* Previous history of 1 or more episodes of ketoacidosis or hyperosmolar state/coma
* Currently receiving chronic (>14 days) systemic glucocorticoid therapy (excluding topical, intraocular, inhaled or intranasal preparations) or have received such therapy within 4 weeks of the screening visit
* Current use of beta-blockers, thiazide diuretic, thyroid products, estrogens, oral contraceptives, phenytoin, nicotinic acid, sympathomimetics, nifedipine and isoniazid and cannot be replaced by any other treatment
* Have any hematologic condition that may interfere with HbA1c measurement (for example, hemolytic anemia, sickle-cell disease)
* Have any other condition (such as, known drug or alcohol abuse or a psychiatric disorder) that may prevent the subject from following and completing the protocol
* Known hypersensitivity to Metformin Hydrochloride
* Currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Any contraindications to Metformin according to local package insert

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., Beijing, China
Locations (1):
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin IR: Subjects received Metformin Immediate Release (IR) tablets, orally once daily (QD) at a dose of 500 milligram (mg) for 1 week, and then the dose was increased with increments of 500 mg every week in the first 2 weeks to 1500 mg. After that, the dose was increased up to a maximum dose of 2000 mg for the next two weeks and maintained at 2000 mg until Week 16.
- Metformin XR: Subjects received Metformin Extended Release (XR) tablets, orally QD at a dose of 500 mg for 1 week, and then the dose was increased with increments of 500 mg every week in the first 2 weeks to 1500 mg. After that, the dose was increased up to a maximum dose of 2000 mg for next 2 weeks and maintained at 2000 mg until Week 16.
Period: Overall Study
Arm/Group | Metformin IR | Metformin XR
Started | 267 | 265
Safety Population | 261 (Out of 261, 12 subjects intolerant to the Metformin IR switched to Metformin XR group.) | 264
Completed | 227 | 222
Not Completed | 40 | 43
Not completed — Adverse Event | 9 | 14
Not completed — Lost to Follow-up | 16 | 8
Not completed — Protocol Violation | 4 | 5
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Other | 4 | 5

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population included all subjects who were randomly allocated to a treatment based on the intention to treat
Groups:
- Metformin IR: Subjects received Metformin IR tablets, orally QD at a dose of 500 milligram (mg) for 1 week, and then the dose was increased with increments of 500 mg every week in the first 2 weeks to 1500 mg. After that, the dose was increased up to a maximum dose of 2000 mg for the next two weeks and maintained at 2000 mg until Week 16.
- Metformin XR: Subjects received Metformin XR tablets, orally QD at a dose of 500 mg for 1 week, and then the dose was increased with increments of 500 mg every week in the first 2 weeks to 1500 mg. After that, the dose was increased up to a maximum dose of 2000 mg for next 2 weeks and maintained at 2000 mg until Week 16.
- Total: Total of all reporting groups
Arm/Group | Metformin IR | Metformin XR | Total
Number analyzed (Participants) | 267 | 265 | 532
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (10.21) | 53.1 (9.72) | 53.8 (9.98)
Gender [Count of Participants; unit: Participants]
  Female | 112 | 108 | 220
  Male | 155 | 157 | 312

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 16
Time Frame: Baseline, Week 16
Population: Per-protocol (PP) population included all subjects who were randomly allocated to a treatment based on intent to treat and were compliant with protocol (absence of any major protocol violations). Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Groups:
- Metformin IR: Subjects received Metformin IR tablets, orally QD at a dose of 500 mg for 1 week, and then the dose was increased with increments of 500 mg every week in the first 2 weeks to 1500 mg. After that, the dose was increased up to a maximum dose of 2000 mg for the next two weeks and maintained at 2000 mg until Week 16.
Arm/Group | Metformin IR | Metformin XR
Number analyzed (Participants) | 208 | 204
Percentage of HbA1c | -1.61 (0.05) | -1.58 (0.05)
Statistical Analysis 1: Comparison: Metformin IR vs Metformin XR; Test type: Non-Inferiority or Equivalence — The non-inferiority margin of this efficacy outcome measure is -0.4%; Least Squares (LS) Mean Difference = 0.03, 95% CI 2-sided [-0.10 to 0.17]

2. Primary Outcome: Overall Gastrointestinal (GI) Tolerability Assessed as Percentage of Subjects With Gastrointestinal Adverse Events During Treatment Period
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Baseline up to Week 16
Population: The safety population included all subjects who received at least 1 dose of trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Metformin IR | Metformin XR
Number analyzed (Participants) | 261 | 264
percentage of subjects | 23.8 [18.72 to 29.39] | 22.3 [17.47 to 27.86]
Statistical Analysis 1: Comparison: Metformin IR vs Metformin XR; Test type: Superiority or Other; p = 0.674, Mantel Haenszel; Percentage difference = -1.52, 95% CI 2-sided [-8.60 to 5.56]

3. Secondary Outcome: Percentage of Subjects With Pre-specified Gastrointestinal Adverse Events During Treatment Period
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. Number of subjects with pre-specified gastrointestinal adverse events (diarrhea, nausea, abdominal pain, bloating, constipation, dyspepsia and flatulence) were reported.
Time Frame: Baseline up to Week 16
Population: The safety population included all subjects who received at least 1 dose of trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Metformin IR | Metformin XR
Number analyzed (Participants) | 261 | 264
percentage of subjects
  Diarrhoea | 16.5 [12.19 to 21.54] | 12.5 [8.76 to 17.10]
  Abdominal Distension | 6.1 [3.54 to 9.76] | 6.4 [3.80 to 10.11]
  Nausea | 6.1 [3.54 to 9.76] | 4.5 [2.37 to 7.81]
  Abdominal Pain | 2.3 [0.85 to 4.94] | 1.9 [0.62 to 4.36]
  Constipation | 1.9 [0.62 to 4.41] | 1.9 [0.62 to 4.36]
  Dyspepsia | 1.1 [0.24 to 3.32] | 0.8 [0.09 to 2.71]
  Flatulence | 0.4 [0.01 to 2.12] | 0 [0.00 to 1.39]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) Level at Week 1, 2, 4, 8, 12 and 16
Time Frame: Baseline, Week 1, 2, 4, 8, 12,16
Population: ITT population included all subjects who were randomly allocated to a treatment based on the intention to treat. Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure. Here "n" signifies those subjects who were evaluable for the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Millimole Per Liter (mmol/L)
Arm/Group | Metformin IR | Metformin XR
Number analyzed (Participants) | 251 | 254
Millimole Per Liter (mmol/L)
  Baseline (n=251, 254) | 8.464 (1.7470) | 8.690 (2.0977)
  Change at Week 1 (n= 249, 248) | -0.647 (1.5615) | -0.736 (1.4305)
  Change at Week 2 (n= 243, 244) | -1.324 (1.4426) | -1.267 (1.9346)
  Change at Week 4 (n= 240, 239) | -1.558 (1.6245) | -1.604 (1.7971)
  Change at Week 8 (n= 219, 230) | -2.075 (1.7359) | -1.999 (2.0192)
  Change at Week 12 (n= 216, 221) | -2.053 (1.7599) | -2.048 (1.8532)
  Change at Week 16 (n= 214, 218) | -1.976 (1.7529) | -2.183 (1.8481)

5. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Plasma Glucose (PPG) Level at Weeks 8 and 16
Description: The 2-hour Postprandial plasma glucose (PPG) level refers to the plasma glucose concentrations after 2 hours of eating.
Time Frame: Baseline, Week 8 and 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Metformin IR | Metformin XR
Number analyzed (Participants) | 223 | 231
mmol/L
  Baseline (n= 223, 231) | 14.604 (3.4334) | 14.764 (3.7705)
  Change at Week 8 (n= 215, 229) | -3.608 (3.6964) | -3.264 (5.9134)
  Change at Week 16 (n= 213, 215) | -3.642 (3.7261) | -3.693 (3.5414)

6. Secondary Outcome: Percentage of Subjects With Hypoglycemia
Description: Hypoglycemia, also called as low blood glucose or low blood sugar, is defined as the blood glucose level of less than normal (that is less than 3.9 millimole per liter [mmol/L]).
Time Frame: Baseline up to Week 16
Population: The safety population included all subjects who received at least 1 dose of trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Metformin IR | Metformin XR
Number analyzed (Participants) | 261 | 264
percentage of subjects | 1.1 [0.24 to 3.32] | 3.0 [1.32 to 5.88]

7. Secondary Outcome: Percentage of Subjects With Marked Hyperglycemia
Description: Marked hyperglycemia was defined as the FPG level of greater than or equal to 11.1 mmol/L.
Time Frame: Baseline up to Week 16
Population: ITT population included all subjects who were randomly allocated to a treatment based on the intention to treat.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Metformin IR | Metformin XR
Number analyzed (Participants) | 267 | 265
percentage of subjects | 0.7 [0.09 to 2.68] | 2.3 [0.84 to 4.86]

8. Secondary Outcome: Percentage of Subjects With HbA1c Less Than (<) 7%
Time Frame: Baseline up to Week 16
Population: ITT population included all subjects who were randomly allocated to a treatment based on the intention to treat.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Metformin IR | Metformin XR
Number analyzed (Participants) | 267 | 265
percentage of subjects | 68.5 [62.60 to 74.06] | 69.8 [63.90 to 75.28]

9. Secondary Outcome: Percentage of Subjects Who Are Totally Intolerant to the Treatment
Description: Subjects were considered to be totally intolerant if they experienced a Grade 3 or higher toxicity considered at least possibly related to the treatment.
Time Frame: Baseline up to Week 16
Population: The safety population included all subjects who received at least 1 dose of trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Metformin IR | Metformin XR
Number analyzed (Participants) | 261 | 264
percentage of subjects | 7.3 [4.44 to 11.13] | 5.7 [3.21 to 9.20]

10. Secondary Outcome: Percentage of Subjects With HbA1c Less Than (<) 7% and With no Severe Gastrointestinal (GI) and Other Adverse Events (AEs)
Description: Percentage of subjects with HbA1c <7% and with no severe GI and other AEs were reported. Severe adverse events were based on Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 and were defined as those events which were medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living (ADL). Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.
Time Frame: Baseline up to Week 16
Population: ITT population included all subjects who were randomly allocated to a treatment based on the intention to treat.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Metformin IR | Metformin XR
Number analyzed (Participants) | 267 | 265
percentage of subjects | 68.2 [62.21 to 73.71] | 69.8 [63.90 to 75.28]

11. Secondary Outcome: Percentage of Subjects Who Are Compliant to Treatment
Description: Compliance was defined as not skipping or forgetting dosing or not delaying the dosing time. Subjects who never missed a dose of medication were considered compliant.
Time Frame: Baseline up to Week 16
Population: The safety population included all subjects who received at least 1 dose of trial treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | Metformin IR | Metformin XR
Number analyzed (Participants) | 261 | 264
percentage of subjects | 99.2 | 99.2

ADVERSE EVENTS:
Time Frame: Baseline up to Week 18
Description: Serious adverse events (SAEs) and Non-SAEs were presented separately for subjects who switched from Metformin IR to Metformin XR group due to intolerance to Metformin IR treatment.
Groups:
- Metformin IR to XR: Subjects who received Metformin IR tablets initially, but were shifted to Metformin XR group due to intolerance to Metformin IR.
Arm/Group | Metformin IR | Metformin XR | Metformin IR to XR
Serious Adverse Events (participants affected / at risk) | 6/249 | 2/264 | 0/12
Other Adverse Events (participants affected / at risk) | 96/249 | 136/264 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin IR (N=249) | Metformin XR (N=264) | Metformin IR to XR (N=12)
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood ketone body increased (Investigations) | 0 | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin IR (N=249) | Metformin XR (N=264) | Metformin IR to XR (N=12)
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Cardiac Discomfort (Cardiac disorders) | 1 | 1 | 0
Palpitations (Cardiac disorders) | 3 | 0 | 0
Right Ventricular Hypertrophy (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Inner Ear Disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Eye Ulcer (Eye disorders) | 0 | 1 | 0
Visual Acuity Reduced (Eye disorders) | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 4 | 9 | 0
Abdominal Distension (Gastrointestinal disorders) | 16 | 17 | 0
Abdominal Pain (Gastrointestinal disorders) | 5 | 5 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 6 | 9 | 1
Abnormal Faeces (Gastrointestinal disorders) | 0 | 3 | 1
Bowel Movement Irregularity (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 5 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 34 | 33 | 9
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Faeces Discoloured (Gastrointestinal disorders) | 0 | 1 | 0
Faeces Hard (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 3 | 9 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 | 4 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 14 | 12 | 3
Vomiting (Gastrointestinal disorders) | 4 | 5 | 0
Asthenia (General disorders) | 2 | 5 | 0
Chest Disconfort (General disorders) | 1 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0
Hangover (General disorders) | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 5 | 8 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 2 | 1 | 0
Periphatic Discomfort (Hepatobiliary disorders) | 0 | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Chronic Hepatitis B (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 4 | 0
Urinary tract Infection (Infections and infestations) | 3 | 9 | 1
Muscle Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 3 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0
Blood Bilirubin increased (Investigations) | 0 | 1 | 0
Blood Glucose Decreased (Investigations) | 1 | 0 | 0
Blood Potassium Decreased (Investigations) | 0 | 1 | 0
Blood Potassium Increased (Investigations) | 0 | 1 | 0
Blood pressure Decreased (Investigations) | 0 | 0 | 1
Blood Sodium Increased (Investigations) | 1 | 0 | 0
Blood Triglycerides Increased (Investigations) | 1 | 0 | 0
Blood uric Acid Increased (Investigations) | 2 | 1 | 0
Electrocardiogram Abnormal (Investigations) | 0 | 1 | 0
Electrocardiogram ST Segment Depression (Investigations) | 1 | 1 | 0
Electrocardiogram ST Segment Elevation (Investigations) | 0 | 1 | 0
Electrocardiogram T Wave Abnormal (Investigations) | 0 | 2 | 0
Electrocardiogram T Wave Amplitude Decreased (Investigations) | 1 | 0 | 0
Gastric PH Decreased (Investigations) | 0 | 1 | 0
Liver Function Test Abnormal (Investigations) | 0 | 1 | 0
Low Density Lipoprotein Increased (Investigations) | 1 | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 1 | 0
Protein Urine Present (Investigations) | 2 | 0 | 0
Urine Ketone Body Present (Investigations) | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 0
White Blood Cell Count Decreased (Investigations) | 1 | 0 | 0
White Blood Cell Count Increased (Investigations) | 0 | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 6 | 5 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 3 | 4 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 5 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 8 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 7 | 11 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Head Discomfort (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 4 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Initial Insomnia (Psychiatric disorders) | 1 | 0 | 0
Libido Decreased (Psychiatric disorders) | 1 | 0 | 0
Listless (Psychiatric disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0
Renal Cyst (Renal and urinary disorders) | 0 | 1 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatic Calcification (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Generalized Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No